CLINICAL TRIAL: NCT00240578
Title: A MULTI-CENTER LONG-TERM FOLLOW-UP STUDY OF PATIENTS WITH LOW-GRADE NON-HODGKIN'S LYMPHOMA PREVIOUSLY TREATED WITH IODINE I 131 TOSITUMOMAB IN STUDIES CP-97-011, CP-98-025, CP-99-032, or CP-99-036
Brief Title: Patients With Low-Grade Non-Hodgkin's Lymphoma Previously Treated With Iodine I 131 Tositumomab
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: BEX104528
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Long-Term Follow-up; BEXXAR; Iodine I 131 Tositumomab; Low-grade lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center study for the long-term follow-up of surviving patients who are expected to complete or who have completed at least two years of follow-up after treatment with Iodine I 131 Tositumomab (BEXXAR) on Studies CP-97-011, CP-98-025, CP-99-032, or CP-99-036. All patients will be assessed for survival and disease status, including subsequent therapy for NHL, and for long-term safety. Additionally Laboratory evaluations consisting of a TSH level and a complete blood cell (CBC) count with a differential and platelet count will be obtained annually. Additionally, patients who remain in long-term response following Iodine I 131 Tositumomab treatment will be followed for response and progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have enrolled in one of the following Corixa sponsored clinical trials: CP-97-011, CP-98-025, CP-99-032, or CP-99-036 and are >2 years post treatment with Iodine I 131 Tositumomab.
* Patients must give written informed consent by signing an IRB/ethics committee approved consent form prior to entry on this follow-up study.

Exclusion Criteria:

* Inability to meet above referenced inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of subjects which have been previously treated with Iodine I 131 Tositumomab in Studies 104505, 93229/023, 393229/007, 104514 and 393229/028.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2003-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
long term followup data | every 3 months at Months 6, 9, 12
  safety and efficacy data will be presented as follow up data with updates to studies 104505, 393229/023, 393229/007, 104514 and 393229/028.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline